CLINICAL TRIAL: NCT04735809
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Assess the Efficacy of a Patented Whole Cell Algae Fermentate on Gut Health in Healthy Adults With Mild Gastrointestinal Issues
Brief Title: Efficacy of a Whole Cell Algae Fermentate on Gut Health and Overall Immune Function in Healthy Adults With Mild Gastrointestinal Issues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kemin Foods LC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: BIO-1901
Record Dates: First submitted 2019-03-27; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2019-03

CONDITIONS: Healthy; Gastrointestinal Dysfunction; Cold Symptom; Flu Symptom

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-Controlled, Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Microcystalline Cellulose
  Interventions: Dietary Supplement: Placebo
- Treatment (Experimental): Whole Cell Algae Fermentate
  Interventions: Dietary Supplement: Whole Cell Algae Fermentate

INTERVENTIONS:
Dietary Supplement: Whole Cell Algae Fermentate — Contains at minimum 50% Beta Glucan
  Arms: Treatment
Dietary Supplement: Placebo — microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The objective of the current study is to evaluate the effect of whole cell fermentate on gut health, including GI system function, such as supporting consistency and regularity of bowel habits, as well as changes in microbiota. The role of the GI system can also be extended to immune regulation because approximately 70% of the entire immune system in the body is located around the gut. Thus, the health and wellbeing of the gut can have a great impact on whole-body health. Therefore, this study will assess the effect on overall immune function.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, crossover trial with a screening visit and two test periods separated by a three-week washout period.

At Visit 1, after subjects have provided informed consent, medical history will be reviewed and clinic visit procedures will be performed, including assessments of prior/current medication/supplement use, and evaluations of inclusion/exclusion criteria.Subjects will be dispensed a diet record, gastrointestinal questionnaire, bowel habits diary, upper respiratory symptom questionnaire, and a stool collection kit to complete prior to Visit 2 (week 0).

At Visit 2 (week 0), eligible subjects will return to the clinic. The stool samples will be collected, and the diet record, gastrointestinal questionnaire, and bowel habits diary will be collected. Subjects will also be administered a stress questionnaire and quality of life questionnaire. Eligible subjects will then be randomized to one of two test groups (placebo or active). Subjects will track study product intake using a daily study product log and track daily cold symptoms. Subjects will also be given a gastrointestinal questionnaire, bowel habits diary, upper respiratory symptom questionnaire, and a stool collection kit to complete prior to Visit 3 (week 4).

At Visit 3 (week 4), the stool samples will be collected, and the diet record, gastrointestinal questionnaire, and bowel habits diary will be collected. Subjects will also be administered a stress and quality of life questionnaire. Unused study product will be collected and compliance assessed via unused study product.Subjects will also be given a gastrointestinal questionnaire, bowel habits diary, and a stool collection kit to complete prior to Visit 4 (week 7)

Subjects will then enter the 3-week washout period, during which time no surveys/questionnaires will be kept and will then crossover to the other study product in their test sequence and repeat the Test Period I procedures (at Visit 2 and 3) during Test Period II (Visits 4 [week 7] and 5 [week 11]).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female, 21-60 years of age
2. Subject has a BMI of 18.5-34.9 kg/m2
3. Subject reports having mild GI issues
4. Subject is willing and able to comply with the collection and storage requirements of the stool samples
5. Subject has internet access via computer, phone or other device and is able to maintain internet access throughout the trial in order to complete online daily questionnaires
6. Subject is a non-user of all tobacco, smoking products and nicotine products
7. Subject is willing to maintain physical activity patterns, body weight, supplements/medications, sleep patterns, and habitual diet throughout the trial.
8. Subject has no health conditions that would prevent him from fulfilling the study requirements 9 Subject understands the study procedures and signs forms providing informed consent to participate in the study

Exclusion Criteria:

1. Subject has an abnormal laboratory test result(s) of clinical importance at Visit 1
2. Subject has a clinically important GI condition that would potentially interfere with the evaluation of the study product
3. Subject has a history or presence of uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including type 1 and type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including unstable depression and/or unstable anxiety disorders) or biliary disorders
4. Subject has a known allergy, intolerance, or sensitivity to any of the ingredients in the study products
5. Subject has extreme dietary habits (e.g., Atkins diet, very high protein, very high fiber)
6. Subject has uncontrolled hypertension
7. Subject has a recent (within 6 weeks of Visit 1) diarrhea (defined as ≥3 loose or liquid stools/d)
8. Subject has participated in colonoscopy or colonoscopy preparation within 3 months prior to Visit 1
9. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer
10. Subject has a history of bariatric surgery for weight reducing purposes
11. Subject has had a weight gain or loss of ≥5% body weight within 6 months of Visit 1
12. Subject has experienced any major trauma or any other surgical event within three months of Visit 1
13. Subject has any signs or symptoms of an active infection (including diarrhea) of clinical relevance within 5 days of Visit 1
14. Subject has used antibiotics within 3 months of Visit 1 or throughout study period
15. Subject has used medications (over-the-counter or prescription) or dietary supplements known to influence GI function
16. Subject has used medications or supplements known to influence immune responses
17. Subject is a regular user (>3 times/week) of prescribed anti-inflammatory medications within 30 d of Visit 1
18. Subject is a regular user (i.e., >1 time per month) of allergy medications
19. Subject has used weight-loss medications
20. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period
21. Subject has a recent history of (within 12 months of screening; Visit 1; week -1) or strong potential for alcohol or substance abuse
22. Individual has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptom | After 4 weeks of each test period
  Gastrointestinal Tolerability Questionnaire
Gastrointestinal ease and consistency | After 4 weeks of each test period
  Bristol Stool Scale
Cold/Flu Symptoms | After 4 weeks of each test period
  Wisconsin Upper Respiratory Symptom Survey

SECONDARY OUTCOMES:
Fecal Microbiome | After 4 weeks of each test period
  Omnigene-GUT DNA Genotek
Fecal biomarker 1 | After 4 weeks of each test period
  Short Chain Fatty Acid
Fecal biomarker 2 | After 4 weeks of each test period
  Leaky Gut biomarker
Stress Questionnaire | After 4 weeks of each test period
  Perceived Stress Questionnaire
Quality of Life Questionnaire | After 4 weeks of each test period
  World Health Organization-Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lawless, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States